CLINICAL TRIAL: NCT01945073
Title: An Educational Intervention to Improve Disease Knowledge Among Adolescents With Sickle Cell Disease
Brief Title: Improving Disease Knowledge in Adolescents With Sickle Cell Disease
Acronym: KNOW-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Monika Parshad-Asnani, Research Fellow, The University of The West Indies
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 0000
Record Dates: First submitted 2013-09-10; First posted 2013-09-18 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Sickle Cell Disease; Quality of Life
Keywords: Educational intervention; Formal Counselling; Knowledge; Illness Perception
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (RC) (No Intervention): Routine clinical care with no intervention
- Educational Booklet (BK) (Experimental): Routine clinical care and educational booklet (BK) given
  Interventions: Behavioral: Educational Booklet (BK)
- Educational Booklet and Counselling (CB) (Experimental): Routine clinical care, aided by formal counselling and active discussions from the educational booklet (CB)
  Interventions: Behavioral: Educational Booklet (BK); Other: Formal Counselling (CB)

INTERVENTIONS:
Behavioral: Educational Booklet (BK) — The information booklet provides age appropriate explanation about SCD: inheritance patterns for the trait and common sickle cell disorders in the Jamaican population. It includes manifestations, complications and the necessary preventive and treatment advice. In addition, issues that are common to adolescents including sexual activity, contraceptive use, drug usage, career advice and developmental changes common to persons with the disease are also discussed.
  Arms: Educational Booklet (BK); Educational Booklet and Counselling (CB)
Other: Formal Counselling (CB) — The study coordinator will have a face to face counselling session, lasting about 30 minutes, with the adolescent and/or caregiver. This will include the use of the educational booklet as an education tool, as well as a thorough discussion on the disease process; its manifestations, effects, and specific concerns during the adolescent period; as well as clarification of common myths and misconceptions about the disease.
  Arms: Educational Booklet and Counselling (CB)

SUMMARY:
Increased knowledge about an illness can increase self-management among those afflicted. In order to facilitate people with sickle cell disease living a longer and healthier life, they should be taught to manage their illness.An adolescent with a chronic illness has many unique challenges, in addition to maneuvering the turbulent adolescence period itself. It has been that better knowledge and more positive perceptions of their illness equate not only to better control of their illness but also better quality of life.Studies have also shown the benefits of self-management: when patients are responsible for managing their own illness, their clinical outcomes and quality of life improve and they become less dependent on health care services.

In this study we aim to examine if knowledge, and any changes in knowledge, will each have any association with Quality of Life (QOL) and their perceptions of their illness (IP). We also seek to investigate the effects of an educational booklet, as well as an intervention including the educational booklet with formal counselling on their knowledge, QOL and IPs.

DETAILED DESCRIPTION:
In this inquiry, we wish to apply an educational intervention to determine if there are any improvements in disease knowledge as a result among adolescents attending the Sickle Cell Unit (SCU) in Jamaica. We also wish to examine if knowledge, and any changes in knowledge, will each have any association with Quality of Life (QOL) and their perceptions of their illness (IP).

Our specific hypotheses are:

1. Important predictors of knowledge among adolescents with Sickle Cell Disease (SCD) are gender, age, education of the adolescent as well as of the parents, socioeconomic status, frequency of attendance at SCU, rural/urban residence, and disease severity.
2. The intervention involving training using an educational booklet specific to 'teens living with SCD' will improve knowledge among the adolescents
3. Adding 'individual Counselling' to the intervention will increase the benefits
4. Improvements in knowledge will translate to improvements in QOL and positive IPs.

ELIGIBILITY:
Inclusion Criteria:

* All adolescent patients, ages 13-19 years inclusive, with Sickle Cell Disease that attend the Sickle Cell Unit at University of the West Indies, Mona Campus will be eligible for the study and hence will be asked to participate.

Exclusion Criteria:

* adolescent with neurological disorders e.g. Cerebrovascular accidents or with physical or intellectual disabilities will be excluded.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Disease Knowledge | 3, 6 and 12 months
  In this inquiry, we wish to apply an educational intervention to determine if there are any improvements in disease knowledge as a result among adolescents attending the Sickle Cell Unit in Jamaica. We also wish to examine if knowledge, and any changes in knowledge, will each have any association with Quality of Life and their perceptions of their illness.

SECONDARY OUTCOMES:
Change in Quality of Life | 3, 6 and 12 months
Change in Illness Perception | 3, 6 and 12 months

OTHER OUTCOMES:
Predictors of change in knowledge | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Monika R Parshad-Asnani, MBBS MSc DM, Principal Investigator — Sickle Cell Unit, TMRI, UWI; Jennifer Knight-Madden, MBBS PhD, Study Director — Sickle Cell Unit, TMRI, UWI
Locations (1):
- Sickle Cell Unit, University of West Indies, Mona Campus, Kingston, Jamaica